CLINICAL TRIAL: NCT02580526
Title: Comparison of Mask Ventilation Techniques in Patients Requiring General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Professor Department of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 150903
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- V-E mask ventilation technique crossover C-E mask ventilation (Active Comparator)
  Interventions: Procedure: V-E mask ventilation for one minute; Procedure: C-E mask ventilation for one minute
- C-E mask ventilation technique crossover V-E mask ventilation (Active Comparator)
  Interventions: Procedure: V-E mask ventilation for one minute; Procedure: C-E mask ventilation for one minute

INTERVENTIONS:
Procedure: V-E mask ventilation for one minute — V-E approach maintains mouth open, creates larger oral cavity and allow positive pressure generated during inspiration to push forwards submandibular region.
  When apnea occurs after anesthesia induction subjects will be ventilated with one of the two techniques randomly, either two-handed "C-E" facemask ventilation technique or with "V-E" technique. Ventilation will be carried out using pressure mode ventilation at respiratory rate of 10 breaths per minute. Subject will start with one technique and then cross over to the other technique.
Procedure: C-E mask ventilation for one minute — Using C-E technique, the operator's fingers pressure mouth closed and push posteriorily the soft tissue of submandibular region.
  When apnea occurs after anesthesia induction subjects will be ventilated with one of the two techniques randomly, either two-handed "C-E" facemask ventilation technique or with "V-E" technique . Ventilation will be carried out using pressure mode ventilation at respiratory rate of 10 breaths per minute. Subject will start with one technique and then cross over to the other technique.

SUMMARY:
This study compares the effectiveness of two kinds of two-handed facemask ventilation techniques (when breathing is supported with machines) at the time that general anesthesia is started. Study participants will start with one technique and then cross over to the other technique.

DETAILED DESCRIPTION:
This study will compare the effectiveness of two-handed V-E mask ventilation technique with the C-E technique. The study hypothesis is based on following considerations:

1. Using C-E technique, the operator's fingers pressure mouth closed and push posteriorily the soft tissue of submandibular region.
2. V-E approach maintains mouth open, creates larger oral cavity and allow positive pressure generated during inspiration to push forwards submandibular region.

Anesthesia care team members, residents or CRNAs familiar with bag-valve mask ventilation, will perform mask ventilation. After receiving preoperative medications, subjects will be placed on the operating table, and electrocardiogram, noninvasive blood pressure, and cutaneous oxyhemoglobin saturation monitoring will be applied. The depth of sedation will be assessed and kept by the care team with IV bolus of propofol.

The sizes of masks will be chosen by the care team and only one size will be used for both techniques. The subject's head will be placed in the neutral position on a pillow and elevate 10 cm from the operating room table, but no backward head tilt or jaw thrust will be performed. One hundred percent oxygen will be delivered throughout the study. The subject will be encouraged to hyperventilate by taking deep breaths to facilitate preoxygenation before the induction of anesthesia.

Pre-oxygenation will be carried out with maximal fresh gas flow and FiO2 1.0 until the expired O2 at or greater than 80%. Then anesthesia will be induced by an intravenous bolus injection of propofol (1-2 mg/kg) after an intravenous bolus injection of fentanyl (50-150 ug).

When the apnea occurs, the subjects will be ventilated with one of the two techniques randomly, either two-handed "C-E" facemask ventilation technique (Group A) or with "V-E" technique (Group B). Ventilation will be carried out using pressure mode ventilation at respiratory rate of 10 breaths per minute, I:E ration of 1:2, peak inspiratory pressure of 20cmH2O and no PEEP. If the expiratory tidal volume is greater than 15ml/kg of ideal body weight, then peak inspiratory pressure will be reduced to 15 cmH2O and 15cm H2O peak inspiratory pressure will be used through the entire the study. The study will be in two steps. Subject will start with one technique (Step 1) and then cross over (Step 2). The subjects in Group A will be first ventilated with "C-E" grip. If the subjects can be adequately ventilated, as defined by perceivable chest movement and carbon dioxide measured during exhalation in the first three breaths, ventilation will continue and complete total 10 breaths (Step 1). Then the subject will be ventilated with two-handed "V-E" grip (Step 2). In Step 1, if the subject cannot be adequately ventilated with C-E grip for even one of the first three breaths, then the subject crosses over and receives V-E grip. If the subject can be adequately ventilated with V-E for at least one of the first 3 breaths, ventilation will continue and complete total 10 breaths. The study will be completed. If the subject cannot be ventilated adequately for at least one of the first three breathes with C-E for the first breaths, nor after crossover with V-E grip, then the study will be terminated and routine care is applied including oral or nasal airway placement, intubation with LMA or tube or waking up the patient.

If subjects are randomized to start with "V-E" technique (Group B), the protocol will be identical to that in Group A except the sequence of applying the two ventilation techniques is reversed.

Upon completion of the study, narcotic and paralytic agent will be given in the usual way and the trachea will be intubated. The oxyhemoglobin saturation will be monitored throughout the study by pulse oximetry and will be maintained > 90%. The study will last about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Requiring general anesthesia in the main operating rooms at Vanderbilt University Medical Center
3. BMI greater than 30

Exclusion Criteria:

1. Untreated ischemic heart diseases
2. Respiratory disorders, including COPD and asthma,
3. American Society of Anesthesiologists (ASA) physical class of 4 or greater,
4. Undergoing emergency surgery,
5. Requiring rapid sequence intubation for aspiration protection,
6. Induction of anesthesia is not done with IV propofol,
7. Requiring fiberoscopic intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-11-17 (Actual)

PRIMARY OUTCOMES:
Difference in expired tidal volume for one minute of each technique | one minute of expired tidal volume for each mask ventilation technique

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheney FW, Posner KL, Lee LA, Caplan RA, Domino KB. Trends in anesthesia-related death and brain damage: A closed claims analysis. Anesthesiology. 2006 Dec;105(6):1081-6. doi: 10.1097/00000542-200612000-00007. PMID 17122570
- [Background] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266
- [Background] Ramachandran SK, Kheterpal S. Difficult mask ventilation: does it matter? Anaesthesia. 2011 Dec;66 Suppl 2:40-4. doi: 10.1111/j.1365-2044.2011.06933.x. PMID 22074078
- [Background] Wong E, Ng YY. The difficult airway in the emergency department. Int J Emerg Med. 2008 Jun;1(2):107-11. doi: 10.1007/s12245-008-0030-6. Epub 2008 May 29. PMID 19384660
- [Background] Orebaugh SL. Difficult airway management in the emergency department. J Emerg Med. 2002 Jan;22(1):31-48. doi: 10.1016/s0736-4679(01)00435-8. PMID 11809554
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity in the United States, 2009-2010. NCHS Data Brief. 2012 Jan;(82):1-8. PMID 22617494
- [Background] Gerstein NS, Carey MC, Braude DA, Tawil I, Petersen TR, Deriy L, Anderson MS. Efficacy of facemask ventilation techniques in novice providers. J Clin Anesth. 2013 May;25(3):193-7. doi: 10.1016/j.jclinane.2012.10.009. Epub 2013 Mar 21. PMID 23523573
- [Derived] Fei M, Blair JL, Rice MJ, Edwards DA, Liang Y, Pilla MA, Shotwell MS, Jiang Y. Comparison of effectiveness of two commonly used two-handed mask ventilation techniques on unconscious apnoeic obese adults. Br J Anaesth. 2017 Apr 1;118(4):618-624. doi: 10.1093/bja/aex035. PMID 28403406